CLINICAL TRIAL: NCT01262781
Title: Is Fructose Linked to Adiposity in Babies?
Acronym: FLAB
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SFGH 6281
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: neonatal adiposity; metabolic syndrome; fructose; maternal diet
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The obesity epidemic has reached down into the infant and toddler age group. Dietary indiscretion during pregnancy, particularly in our current food environment, is a major risk factor for both gestational diabetes and neonatal macrosomia (>4kg newborns), which is itself a risk factor for obesity and metabolic syndrome in the offspring, possibly even during childhood. Temporal increases in fructose consumption in the last two decades coincide with temporal increases weight gain during pregnancy and with increased birth weight, including a higher prevalence of macrosomic newborns. Our central hypothesis is that higher fructose consumption during pregnancy is a risk factor for infant obesity and metabolic syndrome.

DETAILED DESCRIPTION:
The "fetal origins hypothesis" suggests that an individual's risk for obesity and metabolic disorders begins in utero; that fetal or early postnatal exposure to environmental factors, such as maternal nutrition or endocrine disrupting chemicals, adversely influences early development and results in permanent changes affecting energy storage and expenditure.

Most studies on "fetal origins" of obesity in the offspring have focused on maternal high-fat diets; yet dietary fat consumption has not changed appreciably in the last two decades. One chemical exposure in both pregnant mothers and newborns that has been steadily increasing worldwide is fructose. Although ostensibly a carbohydrate, fructose is a potent lipogenic substrate, and in the hypercaloric state, as much as 30% of an ingested fructose load undergoes de novo lipogenesis to form triglyceride thus the effects of high-fat and high-fructose diets in terms of physiology and outcome are comparable. Substituting sucrose (fructose + glucose) for glucose alone increases visceral adiposity, insulin resistance, and dyslipidemia in adult animals and humans. For humans, fructose is ubiquitous in the food environment, especially for pregnant mothers, who are often counseled to drink juice during pregnancy, as it is deemed to be healthier than soda. The effects of fructose consumption during pregnancy on infant birth weight and adiposity has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in all measurements
* Plans to remain in the area through delivery
* Ability to understand and give informed consent in either English or Spanish.

Exclusion Criteria:

* Presence of diabetes prior to the index pregnancy
* Presence of gestational diabetes during a previous pregnancy
* Presence of diabetes or of other chronic metabolic disease such as cardiovascular disease, active thyroid disease, liver disease, pulmonary or psychiatric disorders, HIV
* Any disorder requiring diet therapy (i.e., renal insufficiency)
* Multiple gestation
* Prior history of intrauterine growth retardation
* Use of substances known to cause intrauterine growth retardation (e.g., smoking or drug use). -
* Once recruited, any ultrasonographic evidence of intrauterine growth retardation during the course of the pregnancy would also lead to exclusion.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women between 18 to 40 years of age are eligible for this study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
% adiposity (DEXA) | After delivery, neonatal adiposity will be measured using DEXA. This part of the protocol takes place 4-5 months after recruitment.
  After delivery, neonatal adiposity will be measured using DEXA.

SECONDARY OUTCOMES:
cord blood insulin (corrected by cord blood glucose) | At delivery (in the OR): 4-5 months after recruitment
cord blood triglycerides | At delivery (in the OR): 4-5 months after recruitment
cord blood leptin | At delivery (in the OR): 4-5 months after recruitment
anthropometric measurements on the newborn | After delivery (4-5 months after recruitement)
  birth weight, arm, thigh, and abdominal circumference, subscapular skinfolds
fetal fractional thigh volume obtained by fetal ultrasound | At 32 weeks gestation (4 months after recruitment)
  The fetal fractional thigh volume will me measured in addition to routine fetal measurements at 32 weeks estimated gestation age. This measurement is a measure of neonatal adiposity.
cord blood uric acid | At delivery (in the OR): 4-5 months after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lustig, MD, Principal Investigator — University of California, San Francisco; Anjali Jain, MD, Study Director — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States